CLINICAL TRIAL: NCT01714739
Title: A Phase 1/2 Study of the Combination of Lirilumab (Anti-KIR) Plus Nivolumab (Anti-PD-1) or Lirilumab Plus Nivolumab and Ipilimumab in Advanced Refractory Solid Tumors
Brief Title: A Study of an Anti-KIR Antibody Lirilumab in Combination With an Anti-PD1 Antibody Nivolumab and Nivolumab Plus an Anti-CTLA-4 Ipilimumab Antibody in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA223-001
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: CANCER,NOS
MeSH Terms: conditions — Neoplasms | interventions — lirilumab; Receptors, KIR; Nivolumab; spartalizumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Dose Escalation and Initial Signal Detection in Multiple Solid Tumors - Nivolumab with Lirilumab
  Interventions: Drug: Lirilumab; Drug: Nivolumab
- Part 2 and 3: Cohort Expansion (Experimental): In platinum-refractory recurrent or metastatic SCCHN - Nivolumab with or without Lirilumab
  Interventions: Drug: Lirilumab; Drug: Nivolumab
- Part 4: Cohort Expansion (Experimental): Additional Signal Detection in Solid Tumors - Nivolumab with Lirilumab (Study Part 4 Removed; No Subjects Enrolled)
  Interventions: Drug: Lirilumab; Drug: Nivolumab
- Part 5 and 6 (Experimental): Safety Lead-In and Additional Signal Detection in Solid Tumors -- Nivolumab Plus Ipilimumab with Lirilumab (Study Part 6 Removed; No Subjects Enrolled)
  Interventions: Drug: Lirilumab; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Lirilumab — Specified dose on specified days.
  Other Names: BMS-986015; IPH-2102; ANTI-KIR (Killer-cell Immunoglobulin-like Receptors)
Drug: Nivolumab — Specified dose on specified days.
  Other Names: BMS-936558; ANTI-PD1
Drug: Ipilimumab — Specified dose on specified days.
  Other Names: BMS-734016; Anti-CTLA4
  Arms: Part 5 and 6

SUMMARY:
To assess the safety and tolerability and preliminary anti-tumor activity of lirilumab (BMS-986015) given in combination with nivolumab (BMS-936558) and to identify dose limiting toxicities (DLTs) and the maximally tolerated dose (MTD) of the combination. In addition, to assess the combinations of lirilumab and nivolumab or lirilumab and nivolumab plus ipilimumab (BMS-734016) in subjects with advanced (metastatic and/or unresectable) refractory solid tumors.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* During dose escalation, subjects with advanced solid tumors (except for primary CNS metastases) that have progressed following at least one standard regimen
* During cohort expansion, subjects with various solid tumors that have received at least one and no more than 5 prior treatment regimens
* Subjects must have measurable disease
* Subject must consent to provide previously collected tumor tissue
* Women and men ≥18 years of age with performance status of 0 or 1
* At least 4 weeks since any previous treatment for cancer

Exclusion Criteria:

* Active or chronic autoimmune diseases
* Uncontrolled or significant cardiovascular disease
* Chronic hepatitis (except for subjects with hepatocellular carcinoma)
* Active infection
* Active Central nervous system (CNS) metastases
* Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome((HIV/AIDS)
* Positive test for Hepatitis B virus surface antigen or Hepatitis C antibody (except for subjects with hepatocellular carcinoma)

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2012-10-07 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (30):
- United States (16):
  - Ucsf, San Francisco, California
  - Florida Cancer Affiliates - Ocala, Ocala, Florida
  - University Of Chicago Medical Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Lutherville, Maryland
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Portland Med Ctr, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Eye and Ear Institute, Pittsburgh, Pennsylvania
  - West Cancer Center, Germantown, Tennessee
  - Texas Oncology-Central Austin Cancer Center, Austin, Texas
  - University Of Texas Medical Branch Of Galveston, Galveston, Texas
  - University Of Washington, Seattle, Washington
- Canada (2):
  - Juravinski Cancer Center, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- France (5):
  - Local Institution, Bordeaux
  - Local Institution, Lyon
  - Local Institution, Nice
  - Local Institution, Paris
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - IRCCS Istituto Nazionale Tumori Milano, Milan, MI
  - Local Institution, Siena
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution - 0038, Madrid
  - Local Institution, Madrid
- Switzerland (2):
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 4 and Part 6 of the study were removed from the protocol study design prior to enrolling any subjects.
Groups:
- Part 1/2 Liri 0.1 + Nivo 3: Participants receive Lirilumab 0.1 mg/kg every 4 weeks (Q4W) and Nivolumab 3 mg/kg every 2 weeks (Q2W) for twelve 8-week treatment cycles.
- Part 1/2: Liri 0.3 + Nivo 3: Participants receive Lirilumab 0.3 mg/kg every 4 weeks (Q4W) and Nivolumab 3 mg/kg every 2 weeks (Q2W) for twelve 8-week treatment cycles.
- Part 1/2: Liri 1 + Nivo 3: Participants receive Lirilumab 1 mg/kg every 4 weeks (Q4W) and Nivolumab 3 mg/kg every 2 weeks (Q2W) for twelve 8-week treatment cycles.
- Part 1/2: Liri 3 + Nivo 3: Participants receive Lirilumab 3 mg/kg every 4 weeks (Q4W) and Nivolumab 3 mg/kg every 2 weeks (Q2W) for twelve 8-week treatment cycles.
- Part 3: PBO + Nivo 240: Participants receive Placebo every 4 weeks (Q4W) and a flat dose of nivolumab monotherapy (240mg) every 2 weeks (Q2W) for 8-week cycles until progressive disease.
- Part 3: Liri 240 + Nivo 240: Participants receive Lirilumab 240 mg every 4 weeks (Q4W) and a flat dose of nivolumab 240 mg every 2 weeks (Q2W) for 8-week cycles until progressive disease.
- Part 5: Liri 3 + Nivo 3 + Ipi 1: Participants receive Lirilumab 3 mg/kg IV every 4 weeks (Q4W), Nivolumab 3 mg/kg IV every 2 weeks (Q2W), and Ipilimumab 1 mg/kg IV every 6 weeks (Q6W) for 12-week cycles until progressive disease
Period: Overall Study
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Started | 4 | 16 | 15 | 287 | 2 | 3 | 10
Completed | 0 | 6 | 5 | 23 | 0 | 0 | 0
Not Completed | 4 | 10 | 10 | 264 | 2 | 3 | 10
Not completed — Disease progression | 3 | 5 | 5 | 204 | 1 | 3 | 5
Not completed — Study drug toxicity | 1 | 1 | 1 | 15 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event unrelated to drug | 0 | 0 | 3 | 21 | 0 | 0 | 0
Not completed — Participant request to stop therapy | 0 | 1 | 0 | 6 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 1 | 0 | 8 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 0 | 1 | 1 | 3 | 0 | 0 | 0
Not completed — Poor/non-comliance | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — No longer meets study criteria | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other reason | 0 | 0 | 0 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240 | Part 5: Liri 3 + Nivo 3 + Ipi 1 | Total
Number analyzed (Participants) | 4 | 16 | 15 | 287 | 2 | 3 | 10 | 337
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.3 (12.09) | 58.1 (13.11) | 58.7 (16.85) | 59.7 (11.37) | 65.5 (10.61) | 55.3 (21.08) | 67.1 (10.40) | 59.7 (11.81)
Age, Customized [Count of Participants; unit: Participants] — Age categorical
  Participants
    < 65 years old | 4 | 10 | 9 | 184 | 1 | 2 | 5 | 215
    >= 65 years old | 0 | 6 | 6 | 103 | 1 | 1 | 5 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7 | 80 | 1 | 1 | 1 | 97
  Male | 2 | 11 | 8 | 207 | 1 | 2 | 9 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 4 | 15 | 15 | 175 | 1 | 1 | 8 | 219
  Unknown or Not Reported | 0 | 1 | 0 | 106 | 1 | 2 | 2 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 4 | 16 | 15 | 237 | 2 | 3 | 10 | 287
    Black/African American | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 10
    American Indian / Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Asian | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 10
    Other | 0 | 0 | 0 | 29 | 0 | 0 | 0 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) - Parts 1, 2 and 5
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Parts 1, 2 and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 16 | 15 | 287 | 10
Participants | 4 | 16 | 15 | 284 | 10

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) - Parts 1, 2 and 5
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Parts 1, 2 and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 16 | 15 | 287 | 10
Participants | 1 | 8 | 9 | 205 | 7

3. Primary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation - Parts 1, 2 and 5
Description: Number of participants that experienced an AE leading to discontinuation. An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Parts 1, 2 and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 16 | 15 | 287 | 10
Participants | 1 | 1 | 4 | 49 | 5

4. Primary Outcome: The Number of Participant Deaths in the Study - Parts 1, 2 and 5
Description: The number of participants who died.
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Parts 1, 2 and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 16 | 15 | 287 | 10
Participants | 2 | 7 | 5 | 219 | 5

5. Primary Outcome: Number of Participants With Clinical Laboratory Test Abnormalities - Parts 1, 2 and 5
Description: Number of participants that experienced a clinical laboratory test abnormality, including hematology and serum chemistry, and thyroid panel abnormalities. Abnormalities considered are those Grade 3-4 events with a >= 1 grade increase from baseline. Laboratory tests are graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 where Grade 3 is severe, and Grade 4 is life threatening. Baseline is defined as the last non-missing measurement prior to the first dosing date and time.
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants with available laboratory test measurements. Pre-specified for data to be collected only in Parts 1, 2 and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 16 | 15 | 287 | 10
Participants
  Absolute Neutrophil Count - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 286 | 10
  Absolute Neutrophil Count - Grade 3 | 0 | 0 | 0 | 2 | 0
  Absolute Neutrophil Count - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 286 | 10
  Absolute Neutrophil Count - Grade 4 | 0 | 1 | 0 | 0 | 0
  Alanine Amino Transferase (ALT) - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 277 | 10
  Alanine Amino Transferase (ALT) - Grade 3 | 0 | 0 | 1 | 0 | 0
  Alanine Amino Transferase (ALT) - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 277 | 10
  Alanine Amino Transferase (ALT) - Grade 4 | 0 | 0 | 0 | 0 | 0
  Albumin - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 256 | 2
  Albumin - Grade 3 | 0 | 0 | 0 | 1 | 0
  Albumin - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 256 | 2
  Albumin - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (ALP) - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 277 | 10
  Alkaline Phosphatase (ALP) - Grade 3 | 0 | 1 | 0 | 6 | 0
  Alkaline Phosphatase (ALP) - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 277 | 10
  Alkaline Phosphatase (ALP) - Grade 4 | 0 | 0 | 0 | 0 | 0
  Amylase, Total - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 274 | 8
  Amylase, Total - Grade 3 | 0 | 0 | 0 | 8 | 0
  Amylase, Total - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 274 | 8
  Amylase, Total - Grade 4 | 0 | 0 | 0 | 1 | 0
  APTT - Grade 3: number analyzed (Participants) | 0 | 3 | 1 | 25 | 1
  APTT - Grade 3 |  | 0 | 0 | 0 | 0
  APTT - Grade 4: number analyzed (Participants) | 0 | 3 | 1 | 25 | 1
  APTT - Grade 4 |  | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST) - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 277 | 10
  Aspartate Aminotransferase (AST) - Grade 3 | 0 | 1 | 0 | 4 | 0
  Aspartate Aminotransferase (AST) - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 277 | 10
  Aspartate Aminotransferase (AST) - Grade 4 | 0 | 0 | 1 | 0 | 0
  Bilirubin, Total - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 277 | 10
  Bilirubin, Total - Grade 3 | 0 | 0 | 0 | 1 | 0
  Bilirubin, Total - Grade 4 | 0 | 0 | 0 | 0 | 0
  Calcium, Corrected - Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 61 | 2
  Calcium, Corrected - Grade 3 |  |  |  | 0 | 0
  Calcium, Corrected - Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 61 | 2
  Calcium, Corrected - Grade 4 |  |  |  | 0 | 0
  Calcium, Ionized - Grade 3: number analyzed (Participants) | 0 | 1 | 0 | 2 | 1
  Calcium, Ionized - Grade 3 |  | 0 |  | 0 | 0
  Calcium, Ionized - Grade 4: number analyzed (Participants) | 0 | 1 | 0 | 2 | 1
  Calcium, Ionized - Grade 4 |  | 0 |  | 0 | 0
  Calcium, Total - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 279 | 10
  Calcium, Total - Grade 3 | 0 | 0 | 0 | 6 | 0
  Calcium, Total - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 279 | 10
  Calcium, Total - Grade 4 | 0 | 0 | 0 | 4 | 0
  Creatine Kinase (CK) - Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Creatine Kinase (CK) - Grade 3 |  |  |  | 0 | 0
  Creatine Kinase (CK) - Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Creatine Kinase (CK) - Grade 4 |  |  |  | 0 | 0
  Creatinine - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 278 | 10
  Creatinine - Grade 3 | 0 | 0 | 0 | 0 | 1
  Creatinine - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 278 | 10
  Creatinine - Grade 4 | 0 | 0 | 0 | 0 | 0
  Fibrinogen - Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 47 | 1
  Fibrinogen - Grade 3 |  |  |  | 0 | 0
  Fibrinogen - Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 47 | 1
  Fibrinogen - Grade 4 |  |  |  | 0 | 0
  G-Glutamyl Transferase (GGT) - Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  G-Glutamyl Transferase (GGT) - Grade 3 |  |  |  | 0 |
  G-Glutamyl Transferase (GGT) - Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  G-Glutamyl Transferase (GGT) - Grade 4 |  |  |  | 0 |
  Glucose, Fasting Serum - Grade 3: number analyzed (Participants) | 0 | 1 | 0 | 71 | 2
  Glucose, Fasting Serum - Grade 3 |  | 0 |  | 1 | 0
  Glucose, Fasting Serum - Grade 4: number analyzed (Participants) | 0 | 1 | 0 | 71 | 2
  Glucose, Fasting Serum - Grade 4 |  | 0 |  | 0 | 0
  Glucose, Serum - Grade 3: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Glucose, Serum - Grade 3 |  |  | 0 | 0 |
  Glucose, Serum - Grade 4: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Glucose, Serum - Grade 4 |  |  | 0 | 0 |
  Hemoglobin - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Hemoglobin - Grade 3 | 0 | 1 | 1 | 24 | 1
  Hemoglobin - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Hemoglobin - Grade 4 | 0 | 0 | 0 | 0 | 0
  Leukocytes - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Leukocytes - Grade 3 | 0 | 1 | 0 | 3 | 0
  Leukocytes - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Leukocytes - Grade 4 | 0 | 0 | 0 | 3 | 0
  Lipase, Total (Colorimetric Assay) - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 286 | 10
  Lipase, Total (Colorimetric Assay) - Grade 3 | 0 | 2 | 2 | 18 | 0
  Lipase, Total (Colorimetric Assay) - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 275 | 10
  Lipase, Total (Colorimetric Assay) - Grade 4 | 0 | 0 | 0 | 7 | 0
  Lipase, Total (Turbidimetric Assay) - Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 5 | 0
  Lipase, Total (Turbidimetric Assay) - Grade 3 |  |  |  | 0 |
  Lipase, Total (Turbidimetric Assay) - Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 5 | 0
  Lipase, Total (Turbidimetric Assay) - Grade 4 |  |  |  | 0 |
  Lymphocytes (Absolute) - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Lymphocytes (Absolute) - Grade 3 | 0 | 3 | 4 | 64 | 4
  Lymphocytes (Absolute) - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Lymphocytes (Absolute) - Grade 4 | 0 | 0 | 0 | 9 | 0
  Magnesium, Serum - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 276 | 10
  Magnesium, Serum - Grade 3 | 0 | 0 | 0 | 1 | 0
  Magnesium, Serum - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 276 | 10
  Magnesium, Serum - Grade 4 | 0 | 0 | 0 | 1 | 0
  Neutrophils (Absolute) - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Neutrophils (Absolute) - Grade 3 | 0 | 0 | 0 | 2 | 0
  Neutrophils (Absolute) - Grade 4: number analyzed (Participants) | 0 | 16 | 15 | 281 | 10
  Neutrophils (Absolute) - Grade 4 |  | 1 | 0 | 0 | 0
  pH, Arterial Blood - Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 285 | 0
  pH, Arterial Blood - Grade 3 |  |  |  | 0 |
  pH, Arterial Blood - Grade 4: number analyzed (Participants) | 4 | 0 | 0 | 285 | 0
  pH, Arterial Blood - Grade 4 | 0 |  |  | 0 |
  Phosphorus, Inorganic - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 269 | 10
  Phosphorus, Inorganic - Grade 3 | 0 | 0 | 3 | 10 | 1
  Phosphorus, Inorganic - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 269 | 10
  Phosphorus, Inorganic - Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelet Count - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Platelet Count - Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet Count - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 281 | 10
  Platelet Count - Grade 4 | 0 | 0 | 0 | 1 | 0
  Potassium, Serum - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 278 | 10
  Potassium, Serum - Grade 3 | 0 | 0 | 0 | 6 | 0
  Potassium, Serum - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 278 | 10
  Potassium, Serum - Grade 4 | 0 | 0 | 0 | 3 | 1
  Sodium Serum - Grade 3: number analyzed (Participants) | 4 | 16 | 15 | 278 | 10
  Sodium Serum - Grade 3 | 0 | 1 | 1 | 26 | 1
  Sodium Serum - Grade 4: number analyzed (Participants) | 4 | 16 | 15 | 278 | 10
  Sodium Serum - Grade 4 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the percent of participants whose best overall response (BOR) is either a complete response (CR) or partial response (PR). BOR for a participant was derived using investigator-provided tumor measurements per RECIST v1.1. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose up to approximately 2.5 years
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 16 | 15 | 287 | 2 | 3 | 10
Percentage of participants | 25.0 [0.6 to 80.6] | 37.5 [15.2 to 64.6] | 40.0 [16.3 to 67.7] | 14.6 [10.8 to 19.3] | 50.0 [1.3 to 98.7] | 0 [0.0 to 70.8] | 0 [0.0 to 30.8]

7. Secondary Outcome: Disease Control Rate (DCR) - Part 3
Description: Disease Control Rate (DCR) is defined as the percentage of participants with a best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD). CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. All participants will be monitored by radiographic assessment every 8 weeks from first dose to Week 48, and every 12 weeks thereafter until PD or treatment discontinuation.
Time Frame: From first dose up to approximately 2.5 years
Population: All treated participants. Pre-specified for data to be collected only in Part 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Percentage of participants | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6]

8. Secondary Outcome: Median Duration of Response (mDOR) - Parts 3 and 5
Description: DOR is defined as the time from the date of first response (CR or PR) to the date of first objectively documented tumor progression as determined using RECIST v1.1 or death due to any cause, whichever occurs first. Participant who remain alive and have not progressed were censored on the date of their last evaluable tumor assessment. Participants who started subsequent anticancer therapy without a prior reported progression were censored at the last evaluable tumor assessment prior to initiation of the subsequent anticancer therapy. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose to the date of the first documented tumor progression as determined or death due to any cause, whichever occurs first. (Up to approximately 2.5 years)
Population: All treated participants with a confirmed BOR of CR or PR. Pre-specified for data to be collected only in Parts 3 and 5.
Measure: Median (Full Range); unit: weeks
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 1 | 0 | 0
weeks | NA [40.0 to 40.0] — Insufficient number of participants with events |  |

9. Secondary Outcome: Median Time to Response (mTTR) - Part 3
Description: TTR is defined as the time from the first dosing date to the date of the first documented objective response (CR or PR). CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose of study medication to the date of the first documented objective response (up to approximately 2.5 years)
Population: All treated participants with a confirmed BOR of CR or PR. Pre-specified for data to be collected only in Part 3.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 1 | 0
Weeks | 8.10 [8.1 to 8.1] |

10. Secondary Outcome: The Number of Participants With >=50% or >=80% Tumor Reduction - Parts 3 and 5
Description: Depth of response is defined as the target tumor burden percent change from baseline at nadir for each participant as measured by the number of participants with >= 50% and >= 80% tumor reduction. Tumor assessments are performed every 8 weeks from first dose date for 48 weeks, and then every 12 weeks thereafter until progressive disease (PD) or treatment discontinuation, whichever occurs earlier.
Time Frame: From first dose until progressive disease (PD) or treatment discontinuation, whichever occurs earlier. (Up to approximately 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Parts 3 and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 2 | 3 | 10
Participants
  WITH >=50% TUMOR REDUCTION | 1 | 2 | 0
  WITH >=80% TUMOR REDUCTION | 0 | 1 | 0

11. Secondary Outcome: Overall Survival (OS) - Part 3
Description: Overall Survival (OS) is defined as the time from date of first dose of study medication to the date of death for any cause. A participant who has not died will be censored at last known date alive. OS for a participant who initiated new cancer treatment, will also be censored at the date of the new treatment initiation. Estimated by Kaplan-Meier Method.
Time Frame: From date of first dose of study medication to the date of death for any cause. (Up to approximately 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Part 3.
Measure: Median (Full Range); unit: Years
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Years | NA [0.2 to 1.2] — Time point at which % of survivors drops below 50% has not been reached due to insufficient number of events and/or follow up | 0.3 [0.1 to 0.8]

12. Secondary Outcome: Progression Free Survival (PFS) - Part 3
Description: PFS is defined as the time from the first dosing date to the date of first objectively documented disease progression or death due to any cause, whichever occurs first. Participants who died without a reported prior progression was considered to have progressed on the date of their death. Participants alive with no progression were censored on the last evaluable tumor assessment date. Participants who started subsequent therapy with no prior progression were censored at the last evaluable tumor assessment prior to initiation of the subsequent therapy. Participants with no post-baseline tumor assessment and alive were censored on the date of first dose. Progression is defined as At least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Clinical deterioration in the absence of radiographic evidence is not considered progression.
Time Frame: From first dose to the date of first objectively documented disease progression or death due to any cause, whichever occurs first. (Up to approximately 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Part 3.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Months | NA [1.1 to 11.0] — Insufficient number of events | 1.6 [1.1 to 7.4]

13. Secondary Outcome: Progression Free Survival Rate (PFSR) at 6 Months - Part 3
Description: Percentage of treated participants remaining progression free and surviving at 6 months. For those participants who remain alive and have not progressed, PFS will be censored on the date of the last tumor assessment. Progression is defined as At least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Clinical deterioration in the absence of radiographic evidence is not considered progression.
Time Frame: At 6 months after first dose
Population: All treated participants in Part 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Percentage of participants | 50.0 [0.6 to 91.0] | 33.3 [0.9 to 77.4]

14. Secondary Outcome: Number of Participants With Adverse Events (AEs) - Part 3
Description: as for outcome 1
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Part 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) - Part 3
Description: as for outcome 2
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Part 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

16. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation - Part 3
Description: as for outcome 3
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Part 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

17. Secondary Outcome: The Number of Participant Deaths in the Study - Part 3
Description: The number of participants who died.
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants. Pre-specified for data to be collected only in Part 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Participants | 1 | 3

18. Secondary Outcome: Number of Participants With Clinical Laboratory Test Abnormalities - Part 3
Description: as for outcome 5
Time Frame: From first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years)
Population: All treated participants with available laboratory test measurements. Pre-specified for data to be collected only in Part 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240
Number analyzed (Participants) | 2 | 3
Participants
  Absolute Neutrophil Count - Grade 3 | 0 | 0
  Absolute Neutrophil Count - Grade 4 | 0 | 0
  Alanine Amino Transferase (ALT) - Grade 3 | 0 | 0
  Alanine Amino Transferase (ALT) - Grade 4 | 0 | 0
  Albumin - Grade 3: number analyzed (Participants) | 1 | 1
  Albumin - Grade 3 | 0 | 0
  Albumin - Grade 4: number analyzed (Participants) | 1 | 1
  Albumin - Grade 4 | 0 | 0
  Alkaline Phosphatase (ALP) - Grade 3 | 0 | 0
  Alkaline Phosphatase (ALP) - Grade 4 | 0 | 0
  Amylase, Total - Grade 3: number analyzed (Participants) | 1 | 3
  Amylase, Total - Grade 3 | 1 | 0
  Amylase, Total - Grade 4: number analyzed (Participants) | 1 | 3
  Amylase, Total - Grade 4 | 0 | 0
  APTT - Grade 3: number analyzed (Participants) | 0 | 0
  APTT - Grade 4: number analyzed (Participants) | 0 | 0
  Aspartate Aminotransferase (AST) - Grade 3 | 0 | 0
  Aspartate Aminotransferase (AST) - Grade 4 | 0 | 0
  Bilirubin, Total - Grade 3 | 0 | 0
  Bilirubin, Total - Grade 4 | 0 | 0
  Calcium, Corrected - Grade 3: number analyzed (Participants) | 0 | 2
  Calcium, Corrected - Grade 3 |  | 0
  Calcium, Corrected - Grade 4: number analyzed (Participants) | 0 | 2
  Calcium, Corrected - Grade 4 |  | 0
  Calcium, Ionized - Grade 3: number analyzed (Participants) | 1 | 0
  Calcium, Ionized - Grade 3 | 0 |
  Calcium, Ionized - Grade 4: number analyzed (Participants) | 1 | 0
  Calcium, Ionized - Grade 4 | 0 |
  Calcium, Total - Grade 3 | 0 | 0
  Calcium, Total - Grade 4 | 0 | 0
  Creatine Kinase (CK) - Grade 3: number analyzed (Participants) | 0 | 0
  Creatine Kinase (CK) - Grade 4: number analyzed (Participants) | 0 | 0
  Creatinine - Grade 3 | 0 | 0
  Creatinine - Grade 4 | 0 | 0
  Fibrinogen - Grade 3: number analyzed (Participants) | 0 | 0
  Fibrinogen - Grade 4: number analyzed (Participants) | 0 | 0
  G-Glutamyl Transferase (GGT) - Grade 3 | 0 | 0
  G-Glutamyl Transferase (GGT) - Grade 4: number analyzed (Participants) | 0 | 0
  Glucose, Fasting Serum - Grade 3: number analyzed (Participants) | 0 | 0
  Glucose, Fasting Serum - Grade 4: number analyzed (Participants) | 2 | 2
  Glucose, Fasting Serum - Grade 4 | 0 | 0
  Glucose, Serum - Grade 3: number analyzed (Participants) | 1 | 2
  Glucose, Serum - Grade 3 | 0 | 0
  Glucose, Serum - Grade 4: number analyzed (Participants) | 1 | 3
  Glucose, Serum - Grade 4 | 0 | 0
  Hemoglobin - Grade 3 | 0 | 0
  Hemoglobin - Grade 4 | 0 | 0
  Leukocytes - Grade 3 | 0 | 0
  Leukocytes - Grade 4 | 0 | 0
  Lipase, Total (Colorimetric Assay) - Grade 3 | 0 | 0
  Lipase, Total (Colorimetric Assay) - Grade 4 | 1 | 0
  Lipase, Total (Turbidimetric Assay) - Grade 3: number analyzed (Participants) | 0 | 0
  Lipase, Total (Turbidimetric Assay) - Grade 4: number analyzed (Participants) | 0 | 0
  Lymphocytes (Absolute) - Grade 3 | 0 | 2
  Lymphocytes (Absolute) - Grade 4 | 1 | 0
  Magnesium, Serum - Grade 3 | 0 | 0
  Magnesium, Serum - Grade 4 | 0 | 0
  Neutrophils (Absolute) - Grade 3 | 0 | 0
  Neutrophils (Absolute) - Grade 4 | 0 | 0
  pH, Arterial Blood - Grade 3: number analyzed (Participants) | 0 | 0
  pH, Arterial Blood - Grade 4: number analyzed (Participants) | 0 | 0
  Phosphorus, Inorganic - Grade 3 | 0 | 0
  Phosphorus, Inorganic - Grade 4 | 0 | 0
  Platelet Count - Grade 3 | 0 | 0
  Platelet Count - Grade 4 | 0 | 0
  Potassium, Serum - Grade 3 | 0 | 0
  Potassium, Serum - Grade 4 | 0 | 0
  Sodium Serum - Grade 3 | 0 | 0
  Sodium Serum - Grade 4 | 0 | 0

19. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) - Parts 1, 2 and 5
Description: Number of participants observed as ADA positive at baseline, ADA positive (post-baseline), and ADA negative (post-baseline). Baseline is defined as the last sample before initiation of treatment
  Baseline ADA Positive Participant: A participant with baseline ADA positive sample.
  ADA Positive Participant: Participant with >=1 ADA +ve sample relative to baseline (baseline ADA -ve, or ADA titer >= 9-fold for Lirilumab and >= 4-fold for Nivolumab relative to baseline +ve titer) at any time after first dose during the defined observation time period.
  ADA Negative Participant: A participant with no ADA positive sample after the initiation of treatment.
Time Frame: From first dose to 100 days after last dose (up to approximately 126 weeks)
Population: All participants who receive at least 1 dose of drug and have at least 1 ADA sample available. Pre-specified for data to be collected only in Parts 1, 2, and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 15 | 13 | 255 | 4
Participants
  Baseline ADA Positive - Liri: number analyzed (Participants) | 4 | 11 | 10 | 254 | 4
  Baseline ADA Positive - Liri | 0 | 2 | 0 | 21 | 1
  ADA Positive - Liri: number analyzed (Participants) | 4 | 11 | 10 | 254 | 4
  ADA Positive - Liri | 1 | 1 | 0 | 20 | 0
  ADA Negative - Liri: number analyzed (Participants) | 4 | 11 | 10 | 254 | 4
  ADA Negative - Liri | 3 | 10 | 10 | 234 | 4
  Baseline ADA Positive - Nivo: number analyzed (Participants) | 4 | 15 | 13 | 255 | 3
  Baseline ADA Positive - Nivo | 0 | 1 | 3 | 14 | 1
  ADA Positive - Nivo: number analyzed (Participants) | 4 | 15 | 13 | 255 | 3
  ADA Positive - Nivo | 0 | 1 | 0 | 43 | 0
  ADA Negative - Nivo: number analyzed (Participants) | 4 | 15 | 13 | 255 | 3
  ADA Negative - Nivo | 4 | 14 | 13 | 212 | 3
  Baseline ADA Positive - Ipi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
  Baseline ADA Positive - Ipi |  |  |  |  | 1
  ADA Positive - Ipi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
  ADA Positive - Ipi |  |  |  |  | 0
  ADA Negative - Ipi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
  ADA Negative - Ipi |  |  |  |  | 3

20. Secondary Outcome: The Number of Participants With PD-L1 Status at Pretreatment - Parts 1, 2 and 5
Description: The number of participants with 1% or 5% PD-L1 expression in the tumor cell membrane. Participants are considered positive if they show >=1% or >= 5% PD-L1 expression in the tumor cell membrane and negative if they show < 1% or < 5%. PD-L1 expression is defined as the percent of tumor cells demonstrating plasma membrane PDL1 staining of any intensity. PD-L1 will be evaluated by immunohistochemistry (IHC).
  PD-L1 status at pretreatment is considered positive if any pretreatment sample is positive.
  PDL1= programmed cell death ligand 1
Time Frame: Pre-dose Day 1 (Cycles 1 ,3 ,5, 7, 9), Pre-dose Day 29 (Cycle 1, 2)
Population: All treated participants with available archival tumor sample and with pre- and on-treatment biopsies. Pre-specified for data to be collected only in Parts 1, 2, and 5.
Measure: Number; unit: Number of participants
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 3 | 11 | 13 | 231 | 1
Number of participants
  PD-L1 1 percent - positive | 2 | 5 | 9 | 127 | 1
  PD-L1 1 percent - negative | 1 | 6 | 4 | 104 | 0
  PD-L1 5 percent - positive | 2 | 4 | 4 | 77 | 0
  PD-L1 5 percent - negative | 1 | 7 | 9 | 154 | 1

21. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) - Parts 1, 2 and 5
Description: Pharmacokinetics of lirilumab were derived from serum concentration versus time data. Geometric CV data is not available, therefore the Arithmetic %CV is represented in the table below.
Time Frame: Pre-dose, end of infusion, 24, 168, and 336 hours post dose on day 1 cycle 1 and pre-dose on day 29 cycle 1. Pre-dose, end of infusion, 24 and 168 hours post dose on cycle 2 day 29.
Population: All treated participants who received at least 1 dose of lirilumab and have available serum concentration data. Pre-specified for data to be collected only in Parts 1, 2, and 5.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 13 | 11 | 249 | 2
ng/mL
  Cycle 1 | 2223.10 (NA) — NA = Geometric CV not applicable; %CV = 27 | 6509.35 (NA) — NA = Geometric CV not applicable; %CV = 27 | 22250.96 (NA) — NA = Geometric CV not applicable; %CV = 29 | 52034.18 (NA) — NA = Geometric CV not applicable; %CV = 33 | 65333.91 (NA) — NA = Geometric CV not applicable; %CV = 3
  Cycle 2: number analyzed (Participants) | 3 | 9 | 11 | 111 | 1
  Cycle 2 | 2277.39 (NA) — NA = Geometric CV not applicable; %CV = 6 | 7286.95 (NA) — NA = Geometric CV not applicable; %CV = 24 | 25623.89 (NA) — NA = Geometric CV not applicable; %CV = 20 | 69224.70 (NA) — NA = Geometric CV not applicable; %CV = 26 | 81600.00 (NA) — NA = only 1 participant

22. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] - Parts 1, 2 and 5
Description: as for outcome 21
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 13 | 11 | 249 | 2
hour*ng/mL
  Cycle 1 | 360903.09 (NA) — NA = Geometric CV not applicable; %CV = 23 | 734836.53 (NA) — NA = Geometric CV not applicable; %CV = 45 | 4462883.03 (NA) — NA = Geometric CV not applicable; %CV = 35 | 9647500.52 (NA) — NA = Geometric CV not applicable; %CV = 37 | 8819119.61 (NA) — NA = Geometric CV not applicable; %CV = 29
  Cycle 2: number analyzed (Participants) | 3 | 9 | 11 | 111 | 1
  Cycle 2 | 569516.79 (NA) — NA = Geometric CV not applicable; %CV = 26 | 1367259.80 (NA) — NA = Geometric CV not applicable; %CV = 67 | 6547184.03 (NA) — NA = Geometric CV not applicable; %CV = 37 | 11731186.91 (NA) — NA = Geometric CV not applicable; %CV = 51 | 9958714.89 (NA) — NA = not applicable, only 1 participant

23. Secondary Outcome: Area Under the Plasma Concentration-Time Curve in 1 Dosing Interval [AUC(TAU)] - Parts 1, 2 and 5
Description: as for outcome 21
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 12 | 11 | 209 | 1
hour*ng/mL
  Cycle 1 | 366418.73 (NA) — NA = Geometric CV not applicable; %CV = 21 | 1155363.50 (NA) — NA = Geometric CV not applicable; %CV = 33 | 4462883.03 (NA) — NA = Geometric CV not applicable; %CV = 35 | 11418017.10 (NA) — NA = Geometric CV not applicable; %CV = 28 | 10843715.48 (NA) — NA = not applicable, only 1 participant
  Cycle 2: number analyzed (Participants) | 3 | 6 | 10 | 74 | 0
  Cycle 2 | 569516.79 (NA) — NA = Geometric CV not applicable; %CV = 26 | 1726615.52 (NA) — NA = Geometric CV not applicable; %CV = 44 | 6712959.58 (NA) — NA = Geometric CV not applicable; %CV = 31 | 18504162.18 (NA) — NA = Geometric CV not applicable; %CV = 28 |

24. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) - Parts 1, 2 and 5
Description: Pharmacokinetics of lirilumab were derived from serum concentration versus time data.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 13 | 11 | 249 | 2
hour
  Cycle 1 | 1.13 [1.0 to 1.3] | 1.05 [0.8 to 21.7] | 1.07 [1.0 to 1.6] | 1.22 [0.1 to 161.3] | 1.03 [1.0 to 1.1]
  Cycle 2: number analyzed (Participants) | 3 | 9 | 11 | 111 | 1
  Cycle 2 | 1.08 [1.0 to 1.5] | 1.02 [1.0 to 1.6] | 1.13 [0.9 to 25.5] | 1.18 [0.8 to 168.1] | 1.33 [1.33 to 1.33]

25. Secondary Outcome: Half-life (T-HALF) - Parts 1, 2 and 5
Description: Pharmacokinetics of lirilumab were derived from serum concentration versus time data.
Time Frame: Pre-dose, end of infusion, 24 and 168 hours post dose on cycle 2 day 29.
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 3 | 7 | 7 | 94 | 0
hour | 383.96 (235.421) | 273.89 (234.588) | 515.07 (361.525) | 281.31 (237.236) |

26. Secondary Outcome: Clearance Per Time (CLT) - Parts 1, 2 and 5
Description: as for outcome 21
Time Frame: Pre-dose, end of infusion, 24 and 168 hours post dose on cycle 2 day 29.
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 3 | 6 | 10 | 75 | 0
liter per hour | 0.01 (NA) — NA = Geometric CV not applicable; %CV = 22 | 0.01 (NA) — NA = Geometric CV not applicable; %CV = 38 | 0.01 (NA) — NA = Geometric CV not applicable; %CV = 35 | 0.01 (NA) — NA = Geometric CV not applicable; %CV = 30 |

27. Secondary Outcome: Trough Observed Concentration (Cmin, Also Known as CTAU) - Parts 1, 2 and 5
Description: as for outcome 21
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 12 | 11 | 209 | 1
ng/mL
  Cycle 1 | 87.62 (NA) — NA = Geometric CV not applicable; %CV = 77 | 521.28 (NA) — NA = Geometric CV not applicable; %CV = 60 | 2572.90 (NA) — NA = Geometric CV not applicable; %CV = 47 | 6195.04 (NA) — NA = Geometric CV not applicable; %CV = 45 | 5190.00 (NA) — NA = not applicable, only 1 participant
  Cycle 2: number analyzed (Participants) | 3 | 6 | 10 | 74 | 0
  Cycle 2 | 358.55 (NA) — NA = Geometric CV not applicable; %CV = 68 | 1180.39 (NA) — NA = Geometric CV not applicable; %CV = 65 | 4827.27 (NA) — NA = Geometric CV not applicable; %CV = 32 | 11392.89 (NA) — NA = Geometric CV not applicable; %CV = 45 |

28. Secondary Outcome: Area Under the Pasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time ([AUC(INF)] - Parts 1, 2 and 5
Description: Pharmacokinetics of lirilumab were derived from serum concentration versus time data. AUC(INF) was based on appropriate characterization of the elimination phase of the concentration versus time curve, which was unable to be performed due to limited sampling in this study.
Time Frame: as for outcome 21
Population: All treated participants who received at least 1 dose of lirilumab and have available serum concentration data samples. Due to limited sampling in this study, data was not collected. Pre-specified for data to be collected only in Parts 1, 2, and 5.
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz) - Parts 1, 2 and 5
Description: Pharmacokinetics of lirilumab were derived from serum concentration versus time data. VZ was based on appropriate characterization of the elimination phase of the concentration versus time curve, which was unable to be performed due to limited sampling in this study.
Time Frame: as for outcome 21
Population: as for outcome 28
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: End of Infusion Concentration (Ceoi) - Parts 1, 2 and 5 (Liri)
Description: as for outcome 21
Time Frame: Pre-dose and end of infusion on cycle 1 day 1 and cycle 2 day 29.
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 13 | 11 | 249 | 2
ng/mL
  Cycle 1 Day 1 | 2223.10 (NA) — NA = Geometric CV not applicable; %CV = 27 | 6434.65 (NA) — NA = Geometric CV not applicable; %CV = 28 | 22250.96 (NA) — NA = Geometric CV not applicable; %CV = 29 | 45163.87 (NA) — NA = Geometric CV not applicable; %CV = 38 | 65333.91 (NA) — NA = Geometric CV not applicable; %CV = 3
  Cycle 2 Day 29: number analyzed (Participants) | 3 | 9 | 11 | 110 | 1
  Cycle 2 Day 29 | 2277.39 (NA) — NA = Geometric CV not applicable; %CV = 6 | 7286.95 (NA) — NA = Geometric CV not applicable; %CV = 24 | 25185.06 (NA) — NA = Geometric CV not applicable; %CV = 20 | 65874.20 (NA) — NA = Geometric CV not applicable; %CV = 30 | 81600.00 (NA) — NA = not applicable, only 1 participant

31. Secondary Outcome: Ctrough - Parts 1, 2 and 5 (Liri)
Description: as for outcome 21
Time Frame: Pre-dose on cycle 1 day 29 and Pre-dose and end of infusion on cycle 2 day 29.
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 3 | 12 | 11 | 200 | 1
ng/mL
  Cycle 1 Day 29 | 192.29 (NA) — NA = Geometric CV not applicable; %CV = 42 | 521.28 (NA) — NA = Geometric CV not applicable; %CV = 60 | 2572.90 (NA) — NA = Geometric CV not applicable; %CV = 47 | 6195.08 (NA) — NA = Geometric CV not applicable; %CV = 45 | 5190.00 (NA) — NA = not applicable, only 1 participant
  Cycle 2 Day 29: number analyzed (Participants) | 2 | 9 | 11 | 110 | 1
  Cycle 2 Day 29 | 327.50 (NA) — NA = Geometric CV not applicable; %CV = 85 | 1069.84 (NA) — NA = Geometric CV not applicable; %CV = 63 | 4592.95 (NA) — NA = Geometric CV not applicable; %CV = 32 | 10865.91 (NA) — NA = Geometric CV not applicable; %CV = 45 | 19100.00 (NA) — NA = not applicable, only 1 participant

32. Secondary Outcome: End of Infusion Concentration (Ceoi) - Parts 1, 2 and 5 (Nivo)
Description: Pharmacokinetics of nivolumab were derived from serum concentration versus time data. Geometric CV data is not available, therefore the Arithmetic %CV is represented in the table below.
Time Frame: Pre-dose and end of infusion on cycle 1 day 1 and cycle 2 day 29.
Population: All treated participants who received at least 1 dose of nivolumab and have available serum concentration data. Pre-specified for data to be collected only in Parts 1, 2, and 5.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 15 | 12 | 253 | 6
μg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 15 | 11 | 253 | 6
  Cycle 1 Day 1 | 63.16 (NA) — NA = Geometric CV not applicable; %CV = 31 | 66.33 (NA) — NA = Geometric CV not applicable; %CV = 16 | 66.16 (NA) — NA = Geometric CV not applicable; %CV = 24 | 52.48 (NA) — NA = Geometric CV not applicable; %CV = 25 | 44.75 (NA) — NA = Geometric CV not applicable; %CV = 15
  Cycle 2 Day 29: number analyzed (Participants) | 3 | 9 | 12 | 111 | 2
  Cycle 2 Day 29 | 104.47 (NA) — NA = Geometric CV not applicable; %CV = 16 | 114.89 (NA) — NA = Geometric CV not applicable; %CV = 28 | 116.08 (NA) — NA = Geometric CV not applicable; %CV = 17 | 99.75 (NA) — NA = Geometric CV not applicable; %CV = 25 | 115.37 (NA) — NA = Geometric CV not applicable; %CV = 7

33. Secondary Outcome: Ctrough - Parts 1, 2 and 5 (Nivo)
Description: as for outcome 32
Time Frame: 336 hours post dose on cycle 1 day 1 (cycle 1 day 15) and pre-dose and end of infusion on cycle 2 day 29.
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 5: Liri 3 + Nivo 3 + Ipi 1
Number analyzed (Participants) | 4 | 14 | 15 | 244 | 4
μg/mL
  Cycle 1 Day 15 | 19.15 (NA) — NA = Geometric CV not applicable; %CV = 16 | 20.14 (NA) — NA = Geometric CV not applicable; %CV = 24 | 21.36 (NA) — NA = Geometric CV not applicable; %CV = 24 | 15.81 (NA) — NA = Geometric CV not applicable; %CV = 32 | 17.30 (NA) — NA = Geometric CV not applicable; %CV = 19
  Cycle 2 Day 29: number analyzed (Participants) | 3 | 9 | 13 | 123 | 2
  Cycle 2 Day 29 | 55.67 (NA) — NA = Geometric CV not applicable; %CV = 42 | 62.18 (NA) — NA = Geometric CV not applicable; %CV = 38 | 71.31 (NA) — NA = Geometric CV not applicable; %CV = 21 | 50.07 (NA) — NA = Geometric CV not applicable; %CV = 32 | 62.62 (NA) — NA = Geometric CV not applicable; %CV = 17

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from their first dose until the study was completed (up to approximately 2.5 years). SAEs and Other AEs were assessed from first dose to 150 days post last dose (up to an average of 51 weeks and a maximum of 2.5 years).
Arm/Group | Part 1/2 Liri 0.1 + Nivo 3 | Part 1/2: Liri 0.3 + Nivo 3 | Part 1/2: Liri 1 + Nivo 3 | Part 1/2: Liri 3 + Nivo 3 | Part 3: PBO + Nivo 240 | Part 3: Liri 240 + Nivo 240 | Part 5: Liri 3 + Nivo 3 + Ipi 1
All-Cause Mortality (participants affected / at risk) | 2/4 | 7/16 | 5/15 | 219/287 | 1/2 | 3/3 | 5/10
Serious Adverse Events (participants affected / at risk) | 1/4 | 8/16 | 9/15 | 205/287 | 2/2 | 3/3 | 7/10
Other Adverse Events (participants affected / at risk) | 4/4 | 16/16 | 15/15 | 271/287 | 2/2 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1/2 Liri 0.1 + Nivo 3 (N=4) | Part 1/2: Liri 0.3 + Nivo 3 (N=16) | Part 1/2: Liri 1 + Nivo 3 (N=15) | Part 1/2: Liri 3 + Nivo 3 (N=287) | Part 3: PBO + Nivo 240 (N=2) | Part 3: Liri 240 + Nivo 240 (N=3) | Part 5: Liri 3 + Nivo 3 + Ipi 1 (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 13 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymph node haemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 6 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Salivary gland fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 9 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 14 | 0 | 0 | 0
Secretion discharge (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Actinomycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infective thrombosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 13 | 0 | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 13 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device placement issue (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 13 | 0 | 0 | 0
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 8 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 109 | 1 | 2 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 4 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 24 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 6 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arterial rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1/2 Liri 0.1 + Nivo 3 (N=4) | Part 1/2: Liri 0.3 + Nivo 3 (N=16) | Part 1/2: Liri 1 + Nivo 3 (N=15) | Part 1/2: Liri 3 + Nivo 3 (N=287) | Part 3: PBO + Nivo 240 (N=2) | Part 3: Liri 240 + Nivo 240 (N=3) | Part 5: Liri 3 + Nivo 3 + Ipi 1 (N=10)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 70 | 0 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 8 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 7 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 9 | 0 | 0 | 1
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 7 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 2 | 25 | 1 | 2 | 0
Cataract (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chorioretinal atrophy (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chorioretinal disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Eye movement disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lagophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meibomian gland dysfunction (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Retinal deposits (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 6 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 7 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 10 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 5 | 24 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 9 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 5 | 4 | 60 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 7 | 66 | 0 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1 | 19 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 5 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 29 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 10 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 7 | 62 | 0 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 10 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 5 | 43 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 43 | 0 | 0 | 2
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Chills (General disorders) | 0 | 5 | 1 | 31 | 0 | 0 | 1
Device related thrombosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 15 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 6 | 7 | 144 | 1 | 2 | 3
Influenza like illness (General disorders) | 1 | 0 | 3 | 6 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 5 | 0 | 1 | 1
Malaise (General disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 0
Mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 17 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 9 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 3 | 29 | 0 | 0 | 2
Pain (General disorders) | 0 | 1 | 1 | 8 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 5 | 2 | 69 | 0 | 0 | 1
Swelling face (General disorders) | 0 | 3 | 1 | 2 | 0 | 0 | 1
Xerosis (General disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 11 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Fungal disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital infection fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 7 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 5 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 16 | 1 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 3 | 2 | 7 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 2 | 18 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 5 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 7 | 22 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 13 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 2 | 1 | 19 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 0 | 21 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 13 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 7 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 17 | 0 | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart sounds abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 21 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 5 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Prothrombin time ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 39 | 0 | 3 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 4 | 50 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2 | 17 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 21 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 13 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 9 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 22 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 27 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 28 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 14 | 0 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 8 | 35 | 0 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 34 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 15 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6 | 6 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 9 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 15 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 11 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 26 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 8 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 7 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 3 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 6 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 16 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Consciousness fluctuating (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 4 | 22 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 4 | 44 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 3 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 5 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 2 | 6 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 5 | 7 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 10 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 19 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 8 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 13 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 6 | 15 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 2 | 6 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 6 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulva cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 5 | 62 | 0 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 18 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 47 | 0 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 8 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 10 | 0 | 1 | 0
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4 | 12 | 0 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 7 | 1 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 9 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 11 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 10 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 6 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 5 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 7 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 4 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 12 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 17 | 0 | 0 | 0
Melanocytic hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 6 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 8 | 48 | 0 | 0 | 3
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 7 | 4 | 42 | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 13 | 1 | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 2 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 3 | 0 | 4 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 2 | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 14 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 3 | 19 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT01714739/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT01714739/SAP_001.pdf